CLINICAL TRIAL: NCT03600766
Title: Mirabegron for Treatment of Erectile Dysfunction in Patients With LUTS Secondry to BPH: A Randomized Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MirabegronED
Record Dates: First submitted 2018-07-17; First posted 2018-07-26 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: BPH; Erectile Dysfunction; Prostate Hyperplasia; Erectile Abnormalities; Prostatic Neoplasms
MeSH Terms: conditions — Erectile Dysfunction; Prostatic Hyperplasia; Prostatic Neoplasms | interventions — mirabegron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mirabegron (Active Comparator): oral mirabegron 50 gm plus tamsulosin 0.4 mg once daily for 8 weeks
  Interventions: Drug: Mirabegron
- Placebo (Active Comparator): oral toltordine 4 mg plus tamsulosin 0.4 mg daily for 8 weeks.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Mirabegron — oral mirabegron 50 gm plus tamsulosin 0.4 mg once daily for 8 weeks.
  Arms: Mirabegron
Drug: placebo — oral toltordine 4 mg plus tamsulosin 0.4 mg daily for 8 weeks.
  Arms: Placebo

SUMMARY:
To study the impact of mirabegron, a B3-adrenoceptor agonist, in the treatment of ED in patients with LUTS secondary to BPH and concomitant ED.

DETAILED DESCRIPTION:
Erectile dysfunction (ED) is a major world-wide problem. In United Stated of America, ED affects 26/1000 man yearly (Gonzalgo et al., 2003). The prevalence of ED increases with age from 2-9% in men between 40-49 year, to 20-40% between 60-69 and between 50-100% over 70 years (Gur et al., 2006; Hojanned et al., 2000; Gades et al., 2009; Braun et al., 2000). Many factors may contribute in the occurrence of ED including neuronal, vascular, myogenic and psychological causes (Gur et al., 2016; Johannes et al., 2000, Lewis et al., 2000; Wu et al., 2010; Mallis et al., 2005).

Researchs during the past decade have ﬁrmly established that ED and ejaculatory dysfunction (EJD) are highly prevalent in aging men, particularly those with LUTS of BPH. Furthermore, it has been demonstrated that LUTS of BPH is an independent risk factor for male sexual dysfunction (Hansen BL. et al., 2004).

Although the underlying mechanisms responsible for the relationship between LUTS and male sexual dysfunction are not fully elucidated, possible common links are present including activation of a-adrenergic receptors, endothelial dysfunction, and alterations in sex hormone concentrations and receptor subtypes. Thus, it is now recommended that men presenting with LUTS should be evaluated for sexual dysfunction and those presenting with sexual dysfunction should be evaluated for LUTS (Price DT., et al., 1993).

Also , it is now recognized that certain oral therapies for LUTS/BPH can adversely affect sexual function in patients who are already at increased risk for sexual dysfunction. Moreover, the correction of LUTS was associated with improvement of ED. (De Rose AF., et al., 2002) Healthcare providers should discuss sexual function with BPH patients both before and during treatment. (Raymond C. Rosen et al., 2005) So, use of ED-treating drugs (phosphodiestrase -5 inhibitors) is now a guideline recommendation in the lines of treatment of BPH/LUTS alone or in combination with α blockers. (EUA guidelines, 2015, Gratzke C et., al., 2015).

Phosphodiesterase 5 inhibitors (PDE5i) are effective in treatment of ED. They treat ED through enhancement of the effect of nitric oxide (NO) by inhibition of cyclic guanosin monophosphate (cGMP) breakdown, therefore, increase blood flow through penile arteries. PDE5i are the first-line treatment of ED. Nevertheless, many patients may discontinue the treatment because of side effects, poor response or cost.

It has been shown that B3-adrenoreceptors are mainly localized in the smooth muscle cells of human corpora cavernosa (HCC) (Cirino et al., 2003). The activation of B3-adrenoceptors cause relaxation of the vascular smooth muscle of HCC. Investigators showed that a B3- adrenoreceptors agoinst named "BRL37344" induces relaxation of the HCC. This relaxation has been shown to be linked to inhibition of the RhoA-Rho-associated protein kinase (ROCK) pathway (Cirino et al., 2003). The effect of BRL37344 is mediated by cGMP-dependent but NO-independent mechanisms, altering CC smooth muscle tone and promoting erectile function (Cirino et al., 2003). Thus, b3-adrenoceptor agonists may also serve as potentially useful drugs for the treatment of ED.

Mirabegron is a selective B3-adrenoreceptor agonist and is currently approved in many parts of the world for treatment of overactive bladder (Chapple et al., 2013; Khullar et al., 2013; Chapple et al., 2013; Nitti et al., 2013). Mirabegron displayed 20-200 times higher relative efficacy for human B3-adrenoceptor than that BRL37344 (Takasu et al., 2007). Mirabegron increases intracellular cAMP levels and activates cAMP-dependent protein kinase A resulting in relaxation of the human urinary bladder through a cascade of mechanisms including decrease in intracellular cytoplasmic Ca2+ (Imran et al., 2013; Matanake et al., 2013).

Recently , Gur et al studied the effect of mirabegron on HCC in vitro study and also examined the impact of the drug in vivo, after intracavernosal injection of rats. Authors showed that mirabegron caused marked relaxation of HCC by activating B3-adrenoceptors independently of No pathway. So it appears that mirabegron may be apotential safe and effective therapeutic agent for ED. (Gur et al., 2016) Herein, we designed this protocol to evaluate the role of mirabegron in treating ED in men with BPH/LUTS with concomitant ED.

ELIGIBILITY:
Inclusion Criteria:

* Patients with concomitant ED and irritative LUTS secondary to BPH
* Married and sexually motivated.

Exclusion Criteria:

* Men with Peyronie's disease.
* Patients with contraindication to receive mirabegron (High PVR).
* Psychiatric disorders.
* Previous pelvic surgery or trauma
* Men with prostatic adenocarcinoma
* Patients refusing participating in the study

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male
Enrollment: 50 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
assess change erectile function | 1 year
  measured by International Index of Erectile Function (IIEF).

SECONDARY OUTCOMES:
assess change lower urinary tract symptoms (LUTS) | 1 year
  measured by International Prostate Symptom Score (I-PSS)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Shokeir, PhD, Study Chair — urology and nephrology center
Locations (1):
- Urology and nephrology center, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No